CLINICAL TRIAL: NCT07151326
Title: A Phase II, Single-arm, Multi-center Trial of Cabozantinib for Progressive Hepatocellular Carcinoma (HCC) Post-first-line Immuno-oncologic Combination Therapy (CAPIO Study)
Brief Title: Cabozantinib for Progressive HCC Post-first-line Immuno-oncologic Combination Therapy
Acronym: CAPIO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T 1225; T1225 (Other: TCOG, NHRI)
Record Dates: First submitted 2025-08-14; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Tyrosine kinase inhibitor; Immune checkpoint inhibitor; Multikinase inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): All patients will be treated with cabozantinib at 60 mg once daily.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — All patients will be treated with cabozantinib at 60 mg once daily.
  Other Names: Cabometyx®

SUMMARY:
1. To investigate the efficacy and safety of cabozantinib in patients with progressive HCC after ICI-based combination treatment.
2. To explore potential tissue and peripheral blood biomarkers associated with clinical benefits of cabozantinib, and resistance mechanisms of prior ICI and cabozantinib.

DETAILED DESCRIPTION:
Immune checkpoint inhibitor (ICI)-based combination therapy, such as atezolizumab-bevacizumab or tremelimumab-durvalumab, has become the current standard first-line treatment for advanced hepatocellular carcinoma (HCC). However, there is no approved second-line treatment yet following progression on these ICI-based combination therapies. Multikinase inhibitors (MKIs), such as lenvatinib, sorafenib, cabozantinib, and regorafenib, are often recommended by established guidelines, expert consensus, and retrospective studies. However, this approach lacks robust evidence from prospective studies or reliable biomarkers for patient selection.

Cabozantinib, a MKI targeting vascular endothelial growth factor receptor (VEGFR), MET, and the TAM family of kinases (TYRO3, AXL, and MER), is one of the standard post-sorafenib treatments for advanced HCC. It has shown comparable effectiveness to sorafenib in the first-line setting. The safety profile of cabozantinib is well established and manageable.

Furthermore, cabozantinib offers several advantages that make it a rational treatment option after ICI failure:

1. Potent VEGFR inhibition: Cabozantinib effectively inhibits angiogenesis, which is essential for tumor growth.
2. Additional AXL inhibition: Cabozantinib targets AXL, which is a key mediator of tumor progression and ICI resistance across different cancer types.
3. Clinical evidence: A recent phase II trial demonstrated that around 30% of patients receiving cabozantinib after progression with ICIs remained progression-free at 6 months, despite an objective response rate of 6%. This underscores the need for biomarkers to identify patients who are more likely to benefit from cabozantinib after ICI failure.

In this trial, the investigators aim to investigate the efficacy and safety of cabozantinib in HCC patients who have progressed on first-line ICI-based combination. Additionally, the investigators will explore tumor tissue and peripheral blood biomarkers for clinical benefits of cabozantinib, and resistance mechanisms of prior ICI and current cabozantinib.

ELIGIBILITY:
Inclusion Criteria:

1. Understood and signed the informed consent form
2. Ability to comply with all protocol requirements
3. Age ≥ 18 years when signing informed consent form
4. Diagnosis of HCC confirmed by histology
5. Disease progression following prior first-line ICI-based combination therapy (only atezolizumab plus bevacizumab or tremelimumab plus durvalumab is permitted. Any liver-directed locoregional therapies administered during the treatment period of the first-line ICI-based combination therapy are allowed.
6. Disease that is not amenable to curative surgical and/or locoregional therapies (e.g. surgery, transplant, radiofrequency ablation)
7. At least one measurable target lesion (per RECIST v1.1) that has not been previously treated with local therapy (e.g., radiofrequency ablation, cryoablation, transarterial embolization, transaraterial chemoembolization, radiotherapy, etc.) or, if the target lesion is within the field of previous local therapy, has subsequently progressed in accordance with RECIST v1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Child-Pugh A of liver reserve
10. Adequate hematologic and biochemical profiles:

    * White blood cells (WBC) ≥ 3,000/μL and absolute neutrophil count (ANC) ≥ 1,200/μL without granulocyte colony-stimulating factor support within 1 week before registration
    * Platelets (PLT) ≥ 60,000/μL without transfusion within 1 week before registration
    * Hemoglobin (Hb) ≥ 8 g/dL without transfusion within 1 week before registration
    * Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥ 40 mL/min (using the Cockroft-Gault equation)
    * Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase (ALP) ≤5 × ULN
    * Serum total bilirubin (T-Bil) ≤ 2× ULN
    * Serum albumin (Alb) > 28 g/L (2.8 g/dL)
    * Urinalysis for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours.
11. Recovery to grade 1 from AEs related to any prior treatments, unless the AEs are clinically nonsignificant and/or stable on supportive therapy
12. Subjects with chronic hepatitis B virus (HBV) infection (defined as HBV surface antigen. positive; HBsAg+) must receive antiviral therapy with nucleoside analogs according to the local guidance throughout the study
13. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the study and for 4 months after the last dose of study treatment
14. Life expectancy of 12 weeks or longer

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Prior cabozantinib treatment
3. Any systemic anti-cancer therapy administered after discontinuation of the first-line immune checkpoint inhibitor-based combination
4. Prior liver-directed locoregional therapy administered within 4 weeks before registration
5. Any liver-directed locoregional therapy performed after progression with the first-line immune checkpoint inhibitor-based combination, but palliative radiotherapy for symptomatic bone metastasis is allowed
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before registration
7. Presence of tumor thrombosis or invasion in inferior vena cava (IVC), a major arterial blood vessel (e.g., pulmonary artery or aorta) or heart
8. Subjects with HBV DNA > 2000 IU/mL or detectable hepatitis C virus (HCV) RNA
9. Subjects refuse to provide tumor biopsy specimens within 4 weeks before registration
10. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors.

    (Note: Low dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low dose LMWH (e.g. 40 mg Enoxaparin) for prophylaxis of venous thromboembolism are permitted)
11. Subjects with uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    * Cardiovascular disorders including symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias
    * Uncontrolled hypertension defined as sustained systolic blood pressure (BP) > 150 mm Hg, or diastolic BP > 100 mm Hg despite optimal antihypertensive treatment
    * Stroke (including transient ischemic attack), myocardial infarction, or other ischemic event within 6 months
    * Thromboembolic event within 3 months. (Note: Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumour are eligible)
    * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation/bleeding:
    * Tumours invading the GI tract, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months
12. Major surgery within 2 months before registration. Complete healing from major surgery must have occurred 1 month before registration. Complete healing from minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days before registration
13. Clinically significant bleeding risk including the following within 3 months before registration: upper GI bleeding (including gastroesophageal varices bleeding), hematuria, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
14. Moderate or severe ascites (radiologically detected but clinically insignificant ascites without any diuretics or palliative paracentesis is allowed)
15. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 4weeks before registration (Note: If the QTcF is > 500 ms in first ECG, a total of 3 ECGs should be performed. If the average of these 3 consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility)
16. Previously identified allergy or hypersensitivity to components of the study treatment formulations
17. Inability in swallowing tablets
18. Pregnant or lactating females
19. Diagnosis of another malignancy within 2 years before registration, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
20. Other clinically significant disorders that are judged by investigators to be unsuitable for the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate at 6 months | 30 months
  The percentage of subjects remaining progression (per RECIST v1.1) -free at 6 months after initiation of study treament .
Treatment-emergent adverse event | 30 months
  Incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Study Chair — Taiwan Cooperative Oncology Group, NHRI; Ying-Chun Shen, Principal Investigator — National Taiwan University Hospital
Locations (9):
- Taiwan (9):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital (Lin-Kou),, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Invetigator Initial Trial